CLINICAL TRIAL: NCT03722316
Title: Immersive Nature-based Multimedia Videos to Improve Health in Older Adults With and Without Mild Cognitive Complaints: A Feasibility and Pilot Study.
Brief Title: Nature Video to Improve Older Adult Health: A Feasibility Study.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The presentation of the pandemic made recruitment and implementation impossible for this unfunded study to be completed. We were unable to continue after the loss of key resources.
Sponsor: University of Southern California (Other)
Collaborators: Front Porch Center for Innovation and Wellbeing (Unknown)
Responsible Party: Principal Investigator, Stacey L. Schepens Niemiec, Assistant Professor of Research, University of Southern California
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NatureFeasibility2018
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Mild Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCI/Mild Dementia (Experimental): Twenty participants will be allocated to this arm if they demonstrate mild impairments in cognition based on a cognitive screening phase. Participants enrolled in this arm will be arranged in groups of 5. They will attend a paperwork visit and two video-viewing sessions (order is randomized) held approximately one week apart: (1) brief immersive nature-based video experience + group discussion and (2) comparison condition that includes presentation of a relatively "neutral," un-arousing documentary + group discussion. Each video lasts approximately 15 minutes. Using a semi-structured group discussion guide, participants will be prompted to talk about what they saw in the video and relate video content to their own lives and experiences.
  Interventions: Other: Immersive Nature Video; Other: Neutral Video
- Healthy Older Adults (Active Comparator): Participants are allocated to this arm if they demonstrate healthy cognition based on a cognitive screening phase. Participants enrolled in this arm will be arranged in groups of 5. They will attend a paperwork visit and two video-viewing sessions (order is randomized) held approximately one week apart: (1) brief immersive nature-based video experience + group discussion and (2) comparison condition that includes presentation of a relatively "neutral," un-arousing documentary + group discussion. Each video lasts approximately 15 minutes. Using a semi-structured group discussion guide, participants will be prompted to talk about what they saw in the video and relate video content to their own lives and experiences.
  Interventions: Other: Immersive Nature Video; Other: Neutral Video

INTERVENTIONS:
Other: Immersive Nature Video — An approximately 15-minute digital nature experience using work by filmmaker Louie Schwartzberg-Visual Healing by Moving Art. Time-lapse, high-speed, and macro cinematography are incorporated within each video. Audiovisual content include vivid imagery of a variety of ecosystems and climates accompanied by calming instrumental music.
  Both the MCI/Mild dementia arm and the healthy older adult arm will experience this intervention.
Other: Neutral Video — This video will include clips from relatively non-arousing educational documentaries. Fifteen minutes of documentary content will be selected from a longer video, ensuring that the content remains as neutral as possible. Video selections were modeled after the work from Eryilmaz, Van De Ville, Schwartz, and Vuilleumier (2011) who identified very brief movie clips (i.e., <1 minute) that were rated as neutral as opposed to frightful or enjoyable.
  Both the MCI/Mild dementia arm and the healthy older adult arm will experience this intervention.

SUMMARY:
Background: Exposure to nature has a positive impact on a multitude of health-related outcomes such as stress, attention, recovery after surgery, and overall well-being. There is growing interest in determining the impact of vicarious nature experiences delivered through multimedia platforms on the well-being of persons at high risk for poor psychosocial outcomes, as is the case in older adults diagnosed with mild cognitive impairment (MCI) or mild dementia.

Objectives/Purpose: The primary purpose of this study is to assess the feasibility of providing an immersive nature-based multimedia experience to older adults with MCI or mild dementia. A secondary purpose is to identify the potential health benefits of this intervention.

Methodology: A convenience sample of 40 older adults (65+ years old) with and without mild cognitive complaints will be recruited from a Los Angeles senior service partner. Participation will include three visits. The first visit will include the consent process, cognitive testing, and questionnaire completion. The second and third visits will consist of a video session followed immediately by a group discussion regarding the content in the videos. The two video sessions will be administered in a randomized and counterbalanced manner one week apart. One video involves a 15-minute immersive nature-based experience and the other includes a 15-minute clip that presents emotionally "neutral" educational content. Both sessions will be immediately followed by a group discussion of the content in the videos and how it relates to past experiences.

Outcomes and Analysis: Process evaluation data associated with recruitment, screening eligibility, involvement of personnel, assessment administration, and retention will be collected to determine overall study feasibility. Additionally, selected assessments will be administered at each multimedia experience during key time points to examine potential short-term health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and understands English
* Mild cognitive impairment/mild dementia or normal cognition
* Minor complaints with thinking or memory
* Demonstrate the cognitive capacity to understand and consent to research procedures and to communicate his/her decision

Exclusion Criteria:

* Self-reported phobias that could be triggered by nature-based videos

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Percent of Participants Retained | Initiation of recruitment, through study completion. Average of 6 months.
  The primary outcome of this study is to determine feasibility of study procedures. Retention is one component of feasibility. Retention will be measured as the % completing both video-based visits. Data will be recorded in a testing log.
Recruitment rate | Initiation of recruitment, through study completion. Average of 6 months.
  The primary outcome of this study is to determine feasibility of study procedures. Recruitment rate is one component of feasibility. Recruitment rate will be defined as the % (of number approached) recruited over the duration of the recruitment period. We will also note % recruited from various sources. Data will be recorded in a recruitment log.
Frequency and type of implementation barriers | Initiation of recruitment, through study completion. Average of 6 months.
  The primary outcome of this study is to determine feasibility of study procedures. Implementation barriers is one component of feasibility. Implementation barriers will be defined as the perceived challenges to assessment and intervention delivery on the part of the investigative team. Data sources will include team meeting discussions and study logs made by investigators during implementation.
Number of discussion questions used during group discussion | Day 1 and Day 2 - separated by one week
  The primary outcome of this study is to determine feasibility of study procedures. Intervention fidelity is one component of feasibility. Intervention fidelity will be subjectively determined by adherence to group discussion guides that are paired with the video-based intervention component. Data sources will include video recordings of the group discussion and investigator study notes.

SECONDARY OUTCOMES:
Momentary affective state | Day 1 and Day 2 - separated by one week
  Participants' acute affective state will be assessed using the Multidimensional Mood Questionnaire (MDMQ) - English translation (Steyer, Schwenkmezger, Notz, & Eid, 1994). This 24-item questionnaire addresses degrees of unpleasantness, sleepiness, and restlessness. Items are rated on a 5-point Likert scale ranging from "not at all" to "very much." Subscale items are summed, with higher scores indicated greater well-being.
Working memory | Day 1 and Day 2 - separated by one week
  Working memory will be assessed using a single 2-back test (visual only) administered using a tablet application. In this task, participants will be presented with a digit (0 - 9) that they must temporarily memorize and then indicate if a future stimulus is the same as that digit presented 1 trial previously.
Heart rate variability | Day 1 and Day 2 - separated by one week
  Heart rate will be defined using blood volume pulse signal captured by the E4 empatica wrist monitor.
Skin conductance activity | Day 1 and Day 2 - separated by one week
  Stress/excitement will be defined using skin conductivity changes captured by the E4 empatica wrist monitor.
Quality of social communication | Day 1 and Day 2 - separated by one week
  Video recordings of group discussions will be made to capture social behaviors including communication and interaction. Recordings will subsequently be analyzed using the Holden Communication Scale (Holden & Woods, 1995). This 12-item instrument that addresses factors including conversation, awareness, pleasure, humor, and responsiveness, will be completed by research personnel who will watch and analyze video recordings of each session. Higher scores indicate more impairment with social behavior. The Holden Communication Scale has been determined a valid and reliable assessment for communication ability in persons with dementia (Strøm, Engedal, Benth, & Grov, 2016).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Front Porch Center for Innovation and Wellbeing, Glendale, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided